CLINICAL TRIAL: NCT04148105
Title: Efficacy and Safety of Cilostazol-Nimodipine Combined Therapy on Delayed Cerebral Ischemia After Aneurysmal Subarachnoid Hemorrhage (aSAH): A Prospective, Randomized, Double-Blinded, Placebo-Controlled Trial
Brief Title: Cilostazol and Nimodipine Combined Therapy After Aneurysmal Subarachnoid Hemorrhage (aSAH)
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Insufficient recruitment
Sponsor: Henry Ford Health System (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 1072359
Record Dates: First submitted 2019-10-21; First posted 2019-11-01 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: Aneurysmal Subarachnoid Hemorrhage
Keywords: Delayed cerebral ischemia; Cerebral vasospasm; Cilostazol
MeSH Terms: conditions — Subarachnoid Hemorrhage; Vasospasm, Intracranial | interventions — Cilostazol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): Implement standard treatment regimen of 60 mg nimodipine every 4 hours for 21 days and the standard aneurysmal subarachnoid treatment pathway.
  Interventions: Other: Placebo
- Experimental (Experimental): Administer 100 mg cilostazol, twice daily for 14 days. In addition, implement the standard treatment regimen of 60 mg nimodipine every 4 hours for 21 days, and the standard aneurysmal subarachnoid treatment pathway.
  Interventions: Drug: Cilostazol 100 MG

INTERVENTIONS:
Drug: Cilostazol 100 MG — The addition of 100 mg cilostazol, twice daily for 14 days, to the standard treatment regimen of 60 mg nimodipine every 4 hours for 21 days and the standard aneurysmal subarachnoid treatment pathway
  Arms: Experimental
Other: Placebo — The standard treatment regimen of 60 mg nimodipine every 4 hours for 21 days and the standard aneurysmal subarachnoid treatment pathway
  Arms: Placebo

SUMMARY:
The investigators seek to demonstrate that the combined use of cilostazol and nimodipine will significantly decrease the rate of delayed cerebral infarction and cerebral vasospasm after cerebrovascular intervention when compared to nimodipine alone.

DETAILED DESCRIPTION:
This research study is for people who have a brain hemorrhage, due to a ruptured aneurysm. Adding the drug cilostazol to the standard care may improve outcomes after surgery. The blood within the brain following aneurysmal hemorrhage can have harmful effects on the blood vessels causing them to narrow and thus decrease blood flow; this process is called vasospasm. Decreased blood flow in the brain can lead to more damage. Delayed cerebral ischemia is a complication which is believed to be a consequence of reduced blood flow to the brain following this type of hemorrhage. Cilostazol opens blood vessels and reduces the formation of blood clots. The standard treatment of these hemorrhages currently involves the use of nimodipine which also relaxes blood vessels and allows blood to flow more freely. The combination of these two drugs cilostazol and nimodipine may improve neurologic outcomes after surgery.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Anterior circulation aneurysm
* Patients who have undergone surgical intervention
* Absence of rebleeding or new intracranial hemorrhage noted on post-intervention CT scan
* Consent for study participation

Exclusion Criteria:

* Non-aneurysmal subarachnoid hemorrhage
* Multiple ruptured aneurysms
* Patients with congestive heart failure
* Severe aneurysmal subarachnoid hemorrhage (Hunt Hess Grade V)
* Active pathological bleeding
* Allergy to cilostazol
* Positive pregnancy test
* Coagulopathy not caused by anti-coagulant use
* History of hemorrhagic complications (gastrointestinal bleeding, etc)
* Uncontrolled or severe comorbidity that would qualify as an absolute contraindication for cilostazol
* Patients requiring anticoagulant/antiplatelet treatment following intervention (e.g. stent-assisted coiling or flow-diverting stent obliteration of aneurysm)

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2023-05-21 (Actual); Study Completion 2023-05-26 (Actual)

PRIMARY OUTCOMES:
Delayed Cerebral Infarction | Baseline
  Ischemic lesions demonstrated on follow-up CT or MRI will be interpreted as new cerebral infarctions
Delayed Cerebral Infarction | 1 week (+/- 2 days) postoperatively
  Ischemic lesions demonstrated on follow-up CT or MRI will be interpreted as new cerebral infarctions
Delayed Cerebral Infarction | 1 month (+/- 7 days) postoperatively
  Ischemic lesions demonstrated on follow-up CT or MRI will be interpreted as new cerebral infarctions

SECONDARY OUTCOMES:
Symptomatic Cerebral Vasospasm | At any point leading up to 14 days post-operation
  Development of a new focal or global neurological deficit or deterioration of at least 2 points on the Glasgow Coma Scale which was not explained by initial hemorrhage, re-bleeding, hydrocephalus, surgical complications, fever, infections, or electrolyte or metabolic disturbances; regardless of cerebral infarctions or angiographic vasospasm on imaging
Radiographic Vasospasm | Between 7-10 days postoperatively
  Arterial narrowing not attributable to atherosclerosis, catheter-induced vasospasm, or vessel hypoplasia

OTHER OUTCOMES:
Quality of Life Outcomes: Short-Form 12 | Baseline, 1 month postoperatively, 3 month postoperatively, and 6 month postoperatively
  Short-Form 12 is answered by the patient. On a scale of 0-100, a higher score means better overall physical and mental health.
Modified Rankin Scale | Baseline, 1 month postoperatively, 3 month postoperatively, 6 month postoperatively
  The patient's clinical status is graded on a scale of 0-6. An increasing score means a worse functional outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Boyd Richards, DO, Principal Investigator — Div of Neurosurgery Ascension Providence Hospital MSU College of Human Medicine
Locations (1):
- Ascension Providence Hospital, Southfield, Michigan, United States

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification will be made available following publication upon request at the discretion of the principal investigator.

REFERENCES:
- [Background] D'Souza S. Aneurysmal Subarachnoid Hemorrhage. J Neurosurg Anesthesiol. 2015 Jul;27(3):222-40. doi: 10.1097/ANA.0000000000000130. PMID 25272066
- [Background] Dabus G, Nogueira RG. Current options for the management of aneurysmal subarachnoid hemorrhage-induced cerebral vasospasm: a comprehensive review of the literature. Interv Neurol. 2013 Oct;2(1):30-51. doi: 10.1159/000354755. PMID 25187783
- [Background] Allen GS, Ahn HS, Preziosi TJ, Battye R, Boone SC, Boone SC, Chou SN, Kelly DL, Weir BK, Crabbe RA, Lavik PJ, Rosenbloom SB, Dorsey FC, Ingram CR, Mellits DE, Bertsch LA, Boisvert DP, Hundley MB, Johnson RK, Strom JA, Transou CR. Cerebral arterial spasm--a controlled trial of nimodipine in patients with subarachnoid hemorrhage. N Engl J Med. 1983 Mar 17;308(11):619-24. doi: 10.1056/NEJM198303173081103. PMID 6338383
- [Background] Connolly ES Jr, Rabinstein AA, Carhuapoma JR, Derdeyn CP, Dion J, Higashida RT, Hoh BL, Kirkness CJ, Naidech AM, Ogilvy CS, Patel AB, Thompson BG, Vespa P; American Heart Association Stroke Council; Council on Cardiovascular Radiology and Intervention; Council on Cardiovascular Nursing; Council on Cardiovascular Surgery and Anesthesia; Council on Clinical Cardiology. Guidelines for the management of aneurysmal subarachnoid hemorrhage: a guideline for healthcare professionals from the American Heart Association/american Stroke Association. Stroke. 2012 Jun;43(6):1711-37. doi: 10.1161/STR.0b013e3182587839. Epub 2012 May 3. PMID 22556195
- [Background] Haley EC Jr, Kassell NF, Torner JC. A randomized controlled trial of high-dose intravenous nicardipine in aneurysmal subarachnoid hemorrhage. A report of the Cooperative Aneurysm Study. J Neurosurg. 1993 Apr;78(4):537-47. doi: 10.3171/jns.1993.78.4.0537. PMID 8450326
- [Background] Veldeman M, Hollig A, Clusmann H, Stevanovic A, Rossaint R, Coburn M. Delayed cerebral ischaemia prevention and treatment after aneurysmal subarachnoid haemorrhage: a systematic review. Br J Anaesth. 2016 Jul;117(1):17-40. doi: 10.1093/bja/aew095. Epub 2016 May 8. PMID 27160932
- [Background] Senbokuya N, Kinouchi H, Kanemaru K, Ohashi Y, Fukamachi A, Yagi S, Shimizu T, Furuya K, Uchida M, Takeuchi N, Nakano S, Koizumi H, Kobayashi C, Fukasawa I, Takahashi T, Kuroda K, Nishiyama Y, Yoshioka H, Horikoshi T. Effects of cilostazol on cerebral vasospasm after aneurysmal subarachnoid hemorrhage: a multicenter prospective, randomized, open-label blinded end point trial. J Neurosurg. 2013 Jan;118(1):121-30. doi: 10.3171/2012.9.JNS12492. Epub 2012 Oct 5. PMID 23039152
- [Background] Shibuya M, Suzuki Y, Sugita K, Saito I, Sasaki T, Takakura K, Nagata I, Kikuchi H, Takemae T, Hidaka H, et al. Effect of AT877 on cerebral vasospasm after aneurysmal subarachnoid hemorrhage. Results of a prospective placebo-controlled double-blind trial. J Neurosurg. 1992 Apr;76(4):571-7. doi: 10.3171/jns.1992.76.4.0571. PMID 1545249
- [Background] Dindo D, Demartines N, Clavien PA. Classification of surgical complications: a new proposal with evaluation in a cohort of 6336 patients and results of a survey. Ann Surg. 2004 Aug;240(2):205-13. doi: 10.1097/01.sla.0000133083.54934.ae. PMID 15273542
- [Background] Voldby B, Enevoldsen EM, Jensen FT. Regional CBF, intraventricular pressure, and cerebral metabolism in patients with ruptured intracranial aneurysms. J Neurosurg. 1985 Jan;62(1):48-58. doi: 10.3171/jns.1985.62.1.0048. PMID 3964855
- [Background] Teasdale G, Jennett B. Assessment of coma and impaired consciousness. A practical scale. Lancet. 1974 Jul 13;2(7872):81-4. doi: 10.1016/s0140-6736(74)91639-0. No abstract available. PMID 4136544
- [Background] Frontera JA, Fernandez A, Schmidt JM, Claassen J, Wartenberg KE, Badjatia N, Connolly ES, Mayer SA. Defining vasospasm after subarachnoid hemorrhage: what is the most clinically relevant definition? Stroke. 2009 Jun;40(6):1963-8. doi: 10.1161/STROKEAHA.108.544700. Epub 2009 Apr 9. PMID 19359629
- [Background] Zannad F, Gattis Stough W, McMurray JJ, Remme WJ, Pitt B, Borer JS, Geller NL, Pocock SJ. When to stop a clinical trial early for benefit: lessons learned and future approaches. Circ Heart Fail. 2012 Mar 1;5(2):294-302. doi: 10.1161/CIRCHEARTFAILURE.111.965707. No abstract available. PMID 22438522
- [Background] Puri KS, Suresh KR, Gogtay NJ, Thatte UM. Declaration of Helsinki, 2008: implications for stakeholders in research. J Postgrad Med. 2009 Apr-Jun;55(2):131-4. doi: 10.4103/0022-3859.52846. PMID 19550060
- [Background] Abraham J. International Conference On Harmonisation Of Technical Requirements For Registration Of Pharmaceuticals For Human Use. In: Brouder A, Tietje C, eds. Handbook of Transnational Economic Governance Regimes. Brill 2009. 1041-54. doi:10.1163/ej.9789004163300.i-1081.897
- [Derived] Dawley T, Claus CF, Tong D, Rajamand S, Sigler D, Bahoura M, Garmo L, Soo TM, Kelkar P, Richards B. Efficacy and safety of cilostazol-nimodipine combined therapy on delayed cerebral ischaemia after aneurysmal subarachnoid haemorrhage: a prospective, randomised, double-blinded, placebo-controlled trial protocol. BMJ Open. 2020 Oct 5;10(10):e036217. doi: 10.1136/bmjopen-2019-036217. PMID 33020083